CLINICAL TRIAL: NCT05252949
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial of Oleoylethanolamide (OEA) for Targeting Lipid Metabolism in Gulf War Illness
Brief Title: OEA for Targeting Lipid Metabolism in GWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roskamp Institute Inc. (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RI-OEA-001
Record Dates: First submitted 2022-01-25; First posted 2022-02-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-04

CONDITIONS: Gulf War Illness
MeSH Terms: interventions — oleoylethanolamide

STUDY DESIGN:
Intervention Model Description: We will administer either OEA or placebo to the study participants over a blinded period of 10 weeks, followed by an open label phase with all participants receiving OEA for 5 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Supplement: OEA (Active Comparator): 26 subjects will take the supplement (oleoylethanolamide) during the first phase of the study. 200mg will be taken twice a day for the 10-week period in phase one.
  Interventions: Dietary Supplement: Oleoylethanolamide (OEA)
- Control (Placebo Comparator): 26 subjects will take the placebo during the first phase of the study (10 weeks).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oleoylethanolamide (OEA) — Oleoylethanolamide (OEA) is a naturally occurring ethanolamide that acts as a peroxisome proliferator-activated receptor alpha (PPAR-α) agonist, thereby modulating lipid profiles.
  Arms: Study Supplement: OEA
Dietary Supplement: Placebo — Visually matching placebo capsules will contain the same inactive ingredients present in the manufactured OEA capsules, with the exception of any OEA compound.
  Arms: Control

SUMMARY:
The study is a single site, randomized, double-blind, placebo-controlled study with an open label extension to evaluate the effects of Oleoylethanolamine (OEA) on blood lipid and immune biomarkers in participants with Gulf War Illness (GWI).

DETAILED DESCRIPTION:
The 1991 Gulf War (GW) was fought by a coalition of 30 countries that included 700,000 U.S. troops. Although the war itself lasted two months, adverse health consequences from this conflict are still experienced by GW veterans. Soon after their return, many soldiers started reporting multiple, seemingly unrelated symptoms, such as memory impairment, fatigue, gastrointestinal problems, and widespread pain. This illness is termed Gulf War Illness (GWI) and affects about 32% of GW veterans. Several animal studies suggest that GWI presentation involves disturbed immune responses in the brain that correspond with altered lipid metabolism. Many of these lipid alterations are detected in blood of veterans with GWI and point to an abnormal function of peroxisomes and mitochondria which regulate lipids that are required for cellular signaling and for maintaining normal physiology. The investigators' preclinical studies using a GWI mouse model showed that targeting peroxisomal lipid metabolism with oleoylethanolamide (OEA) reduced corrected immune function and normalized brain and blood lipid profiles in GWI mice. Therefore, the objective of this pilot clinical research study is to determine if OEA supplementation in veterans with GWI maintains healthy blood lipid and immune profiles.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, all ethnic groups, and ages up to 70.
* Subject willing and able to give informed consent.
* Medically stable as per the investigator's discretion.
* Negative urine pregnancy test for females of childbearing potential. A woman is considered of childbearing potential unless she is surgically sterile (hysterectomy or tubal ligation) or is postmenopausal (no menstrual cycle for 2 years or more).
* Must be willing to use adequate birth control during the study and for 30 days after the last dose. Females agreeing to take an acceptable form of birth control per investigator discretion (where relevant). Females must prevent pregnancy or otherwise be unable to conceive.
* Veterans deployed to the Gulf War between August 1990 and August 1991.
* Veteran meets criteria for the CDC Chronic Multisymptom Illness (CMI) GWI definition or Kansas GWI definition.
* Weight of 50.0kg - 200.0kg (110lbs - 440lbs).

Exclusion Criteria:

* Diagnosed by a physician with medical or psychiatric conditions that would account for their symptoms or interfere with their ability to report their symptoms.
* Female subject is either pregnant or nursing.
* Have contraindications, allergy, or sensitivity to OEA, olive oil, or excipients (microcrystalline cellulose, silicon dioxide, magnesium stearate, macrogol polyvinyl alcohol copolymer, talc, titanium dioxide, glycerol monocaprylocaprate and polyvinyl alcohol).
* Any significant medical condition that could interfere with study conduct, as per investigator discretion. These may include but are not limited to the following: untreated chronic hypertension (defined as systolic > 180 mmHg; diastolic >110 mmHg), myocardial infarction within 6 months of screening, renal failure, hepatic failure, and/or receiving chemotherapy.
* Clinically significant lab values for clinical laboratory assessments.
* Poor venous access.
* Current use of any OEA supplement products within 30 days of screening.
* Participation in another clinical trial involving dietary or pharmaceutical intervention within 90 days of screening.

Max Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Changes in lipid biomarker profiles | 10 weeks
  The primary objective of the study is to assess the change in lipid levels in the blood between the two treatment arms over the 10-week placebo-controlled phase.
Changes in immune biomarker profiles | 10 weeks
  The primary objective of the study is to assess the change in cytokine levels in the blood between the two treatment arms over the 10-week placebo-controlled phase.

SECONDARY OUTCOMES:
Changes in fatigue | 10 weeks
  The study will use the Multidimensional Fatigue Inventory (MFI-20) to assess fatigue.
Changes in mood | 10 weeks
  The study will use the Profile of Mood States (POMS) to assess mood.
Changes in pain | 10 weeks
  The study will use the McGill Pain Questionnaire (SF-MPQ) to assess pain.
Changes in cognition (neurocognitive) | 10 weeks
  The study will use the CNS Vital Signs computerized neurocognitive assessment software to assess memory. The computerized test uses individual tests to comprise a neurocognitive index score that can be used to evaluate neurocognitive status.
Changes in cognition (neuropsychological) | 10 weeks
  The study will use the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) cognitive test to assess memory. The test incorporates immediate memory, visuospatial/constructional, language, attention, and delayed memory components to determine a total scaled score for neuropsychological status. This total score ranges from 200 to 800, with higher scores increasing the associated percentile.
Changes in quality of life | 10 weeks
  The study will use the Quality of Life Scale (SF36).

CONTACTS AND LOCATIONS:
Overall Officials: Laila Abdullah, PhD, Principal Investigator — The Roskamp Institute; Michael Hoffmann, MD, Principal Investigator — The Roskamp Institute
Locations (1):
- The Roskamp Institute, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White RF, Steele L, O'Callaghan JP, Sullivan K, Binns JH, Golomb BA, Bloom FE, Bunker JA, Crawford F, Graves JC, Hardie A, Klimas N, Knox M, Meggs WJ, Melling J, Philbert MA, Grashow R. Recent research on Gulf War illness and other health problems in veterans of the 1991 Gulf War: Effects of toxicant exposures during deployment. Cortex. 2016 Jan;74:449-75. doi: 10.1016/j.cortex.2015.08.022. Epub 2015 Sep 25. PMID 26493934
- [Background] Abdullah L, Crynen G, Reed J, Bishop A, Phillips J, Ferguson S, Mouzon B, Mullan M, Mathura V, Mullan M, Ait-Ghezala G, Crawford F. Proteomic CNS profile of delayed cognitive impairment in mice exposed to Gulf War agents. Neuromolecular Med. 2011 Dec;13(4):275-88. doi: 10.1007/s12017-011-8160-z. Epub 2011 Oct 11. PMID 21986894
- [Background] Abdullah L, Evans JE, Bishop A, Reed JM, Crynen G, Phillips J, Pelot R, Mullan MA, Ferro A, Mullan CM, Mullan MJ, Ait-Ghezala G, Crawford FC. Lipidomic profiling of phosphocholine-containing brain lipids in mice with sensorimotor deficits and anxiety-like features after exposure to Gulf War agents. Neuromolecular Med. 2012 Dec;14(4):349-61. doi: 10.1007/s12017-012-8192-z. Epub 2012 Jul 14. PMID 22798222
- [Background] Abdullah L, Evans JE, Montague H, Reed JM, Moser A, Crynen G, Gonzalez A, Zakirova Z, Ross I, Mullan C, Mullan M, Ait-Ghezala G, Crawford F. Chronic elevation of phosphocholine containing lipids in mice exposed to Gulf War agents pyridostigmine bromide and permethrin. Neurotoxicol Teratol. 2013 Nov-Dec;40:74-84. doi: 10.1016/j.ntt.2013.10.002. Epub 2013 Oct 17. PMID 24140745
- [Background] Abdullah L, Evans JE, Joshi U, Crynen G, Reed J, Mouzon B, Baumann S, Montague H, Zakirova Z, Emmerich T, Bachmeier C, Klimas N, Sullivan K, Mullan M, Ait-Ghezala G, Crawford F. Translational potential of long-term decreases in mitochondrial lipids in a mouse model of Gulf War Illness. Toxicology. 2016 Nov 30;372:22-33. doi: 10.1016/j.tox.2016.10.012. Epub 2016 Oct 29. PMID 27931520
- [Background] Joshi U, Evans JE, Joseph R, Emmerich T, Saltiel N, Lungmus C, Oberlin S, Langlois H, Ojo J, Mouzon B, Paris D, Mullan M, Jin C, Klimas N, Sullivan K, Crawford F, Abdullah L. Oleoylethanolamide treatment reduces neurobehavioral deficits and brain pathology in a mouse model of Gulf War Illness. Sci Rep. 2018 Aug 27;8(1):12921. doi: 10.1038/s41598-018-31242-7. PMID 30150699
- [Background] Emmerich T, Zakirova Z, Klimas N, Sullivan K, Shetty AK, Evans JE, Ait-Ghezala G, Laco GS, Hattiangady B, Shetty GA, Mullan M, Crynen G, Abdullah L, Crawford F. Phospholipid profiling of plasma from GW veterans and rodent models to identify potential biomarkers of Gulf War Illness. PLoS One. 2017 Apr 28;12(4):e0176634. doi: 10.1371/journal.pone.0176634. eCollection 2017. PMID 28453542
- [Derived] Abdullah L, Keegan AP, Hoffmann M, Baraniuk J, Mack W, Sullivan K, Luis C, Rindfleisch C, Huguenard CJC, Cseresznye A, Aldrich GJ, Evans JE, Paris D, Helgager D, Crawford F, Mullan M. Oleoylethanolamide supplementation improves mood and reduces fatigue in veterans with GWI in a 15-week randomized, double-blind, placebo-controlled exploratory clinical trial. Sci Rep. 2026 Jan 9;16(1):4933. doi: 10.1038/s41598-026-35168-3. PMID 41513981